CLINICAL TRIAL: NCT07191977
Title: Neoadjuvant Camrelizumab With Palbociclib for the Treatment of Resectable Esophageal Squamous Cell Carcinoma: A Single-Arm Phase 2 Trial
Brief Title: Neoadjuvant Camrelizumab With Palbociclib for Resectable Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-417
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Squamour Cell Cancer
MeSH Terms: interventions — camrelizumab; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab+Palbociclib(100mg) (Experimental)
  Interventions: Drug: Camrelizumab; Drug: Palbociclib

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab will be given at at a dose of 200 mg intravenously on day 23 of a planned 28-day cycle, and two doses before surgery.
Drug: Palbociclib — Palbociclib will be given at a dose of 100 mg every day orally with three weeks on and one week off. Four weeks is a cycle and it will be given for three cycles.

SUMMARY:
The goal of this Phase 2 clinical trial is to learn if the combination of Camrelizumab and Palbociclib is a safe and effective treatment when given before surgery (neoadjuvant therapy) for patients with esophageal squamous cell carcinoma (ESCC) that can be surgically removed. Camrelizumab is an immunotherapy drug that helps the immune system fight cancer, and Palbociclib is a targeted therapy drug that stops cancer cells from growing.

The main questions it aims to answer are:

Is the combination of Camrelizumab and Palbociclib safe for patients to receive before their surgery? How effective is this treatment combination in shrinking tumors prior to surgery?

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with esophageal squamous cell cancer by gastroscopic biopsies.
* The primary tumor should be located in the thorax and evaluated resectable( cT1b-T3N1-3M0, cT3N0M0) by CT/MRI/EUS
* The patients should be at the range of 18-75 years old, Eastern Cooperative Oncology Group (ECOG) 0-1.
* The patients should have no functional disorders in major organs. Blood routine tests, as well as lung, liver, kidney, and heart functions should be basically normal.
* The patients should be able to understand our research and be willing to accept surgical treatment and sign the informed consent.

Exclusion Criteria:

* The stage of tumor is T4b (AJCC/International Union Against Cancer (UICC) 8th Edition) and cannot be resected.
* Currently undergoing other chemotherapy, radiotherapy, targeted therapy or immunotherapy.
* History of other malignancies.
* Have an active autoimmune disease requiring systemic treatment or a documented history of clinically severe autoimmune disease.
* Any history of allergic disease, or a sever hypersensitivity reaction to drugs, or allergy to the study drug components.
* Presence of serious medical diseases, such as grade II and above cardiac dysfunction (NYHA criteria), ischemic heart diseases, etc.
* The patients with severe systematic intercurrent diseases, including active infection or poorly controlled diabetes, coagulation disorders, hemorrhagic tendency, or those undergoing thrombolysis or anticoagulant therapy etc. are excluded from the study.
* Female participants who test positive for a serum pregnancy test, are in the lactation period, or are at a childbearing stage and unwilling to use contraception measures during the research are excluded.
* Received any investigational drug within 4 weeks prior to the first dose, or concurrently enrolled in another clinical trial.
* Any other factors that are not suitable for inclusion in this study judged by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Major Pathologic Response | up to 15 weeks
  Major Pathologic Response (MPR) was defined as fewer than 10% viable tumor cells.

SECONDARY OUTCOMES:
Pathological Complete Response (PCR) | up to 15 weeks
  The pCR will be defined as the proportion of participants with absence of residual tumor in the resected primary tumor and all resected lymph nodes after completion of neoadjuvant treatment.
Overall survival (OS) | Up to 2 years
  Proportion of participants who achieve survival post treatment
Objective response rate (ORR) | up to 15 weeks
  Proportion of participants with measurable disease at baseline and have been re-evaluated after at least 1 cycle of therapy with observed reduction in tumor burden as defined by RECIST and iRECIST criteria after 2 doses of Proportion of participants with measurable disease at baseline and have been re-evaluated after at least 1 cycle of therapy with observed reduction in tumor burden as defined by RECIST and iRECIST criteria after 2 doses of camrelizumab and palbociclib
R0 resection rate | up to 15 weeks
  This will be defined as the proportion of participants with R0 resection
Incidence of Treatment-Emergent Adverse Events | from the first dose to within 30 days after the last dose
  Number of participants who experience grade 1 or higher adverse events, as defined by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Zhou, Principal Investigator — West China Hospital